CLINICAL TRIAL: NCT04500483
Title: Measurement of Resting Energy Expenditure in Burn or Critically Ill Patients at Risk of Malnutrition
Brief Title: Indirect Calorimetry in Patients at Risk of Malnutrition
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of clinic, University of Liege
Other Study IDs: CaloIF
Record Dates: First submitted 2020-08-01; First posted 2020-08-05 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Burns; Critical Illness; Indirect Calorimetry; Resting Energy Expenditure; Nutrition Disorders
MeSH Terms: conditions — Burns; Critical Illness; Nutrition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Burn outpatients: Burn patients treated for minor burns in an outpatient setting
  Interventions: Diagnostic Test: indirect calorimetry
- ICU survivors: Critically ill patients who survived ICU stay and are admitted in a general ward
  Interventions: Diagnostic Test: indirect calorimetry

INTERVENTIONS:
Diagnostic Test: indirect calorimetry — measurement of resting energy expenditure using indirect calorimetry

SUMMARY:
Burn patients treated in an outpatient clinic and ICU survivors are at risk of malnutrition. There are no clear guidelines determining the energy target in those two populations. The aim of this observation study is to measure the resting energy expenditure of those patients, using indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* minor burn treated in an outpatient setting
* ICU survivor, who was discharged from ICU after a stay of at least 7 days

Exclusion Criteria:

* oxygen supply
* chest drainage
* not french speaking
* confusion, coma
* cognitive disorder
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the study population is divided into two groups: burn patients with minor burn exclusively treated in an outpatient setting, and ICU survivors who were discharged fro ICU after a stay of at least 7 days
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
resting energy expenditure | during the 7 days following injury in burn patients or following ICU discharge in ICU survivors

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No